CLINICAL TRIAL: NCT00729196
Title: A Trial of Two Diets for Weight and Diabetes Management
Acronym: Two-for-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Anthony N. Fabricatore, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23 DK70777 (completed); K23DK070777 (NIH)
Record Dates: First submitted 2008-08-05; First posted 2008-08-07 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: Obesity; Type 2 Diabetes; Glycemic Load; Weight Loss; Glycated Hemoglobin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Low-Glycemic Load Diet
  Interventions: Behavioral: Lifestyle Modification
- 2 (Active Comparator): Low-Fat Diet
  Interventions: Behavioral: Lifestyle Modification

INTERVENTIONS:
Behavioral: Lifestyle Modification — Weekly group therapy for 20 weeks, followed by bi-weekly group therapy for 20 weeks

SUMMARY:
The purpose of this study is to determine whether a low-fat or low-glycemic load diet is more effective for controlling weight and blood glucose in persons with type 2 diabetes.

DETAILED DESCRIPTION:
This research is a randomized controlled trial to compare long-term outcomes behavioral weight loss interventions that include either low-fat or low-glycemic load dietary instruction. Targets for energy intake and expenditure, and behavioral skills taught, are identical across the two diets. Additionally, both treatments include 20 weekly group sessions, followed by 10 every-other-week sessions. Participants are overweight and obese adults with type 2 diabetes. The primary outcomes are changes in weight and glycated hemoglobin. Those randomized to the low-glycemic load diet are expected to achieve greater weight losses and maintain better glycemic control at the end of treatment (i.e., week 40) and after 1 year of no-treatment follow-up (i.e., week 92).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Body mass index (BMI) of 27 to 45 kg/m2 with weight </= 136 kg (300 lbs.
* Capacity to provide written informed consent
* Systolic blood pressure between 90 and 160 mm Hg, inclusive.
* Diastolic blood pressure between 65 and 100 mm Hg, inclusive.
* Resting heart rate between 65 and 90 beats per minute, inclusive.

Exclusion Criteria:

* a recent (i.e., within 1 year) myocardial infarction
* unstable angina
* malignant arrhythmias
* history of cerebrovascular, renal, or hepatic disease
* history of seizures
* protein wasting diseases (e.g., Cushing's syndrome)
* uncontrolled hypertension (> 160/100 mm Hg)
* type 1 diabetes
* uncontrolled thyroid disease
* pregnancy or lactation
* electrolyte abnormalities
* clinically significant psychosocial impairment (principally, major depression)
* treatment with steroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-07; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Percent change in weight | 92 weeks

SECONDARY OUTCOMES:
Change in HbA1c | 92 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anthony N Fabricatore, Ph.D., Principal Investigator — University of Pennsylvania; Thomas A Wadden, Ph.D., Study Director — University of Pennsylvania; Virginia A Stallings, M.D., Study Director — Children's Hospital of Philadelphia; Stanley Schwartz, M.D., Study Director — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States